CLINICAL TRIAL: NCT06464705
Title: Effect of Pulsed Electromagnetic Fields on Promoting Hamstring Muscle Strength After Anterior Cruciate Ligament Reconstruction With Hamstring Autograft: A Double-Blind, Placebo-Controlled, Randomised Clinical Trial
Brief Title: To Investigate the Effect of PEMF for Pateitns After Anterior Cruciate Ligament Reconstruction With Hamstring Autograft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Pauline Lui, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.130
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Hamstring Muscle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMF treatment (Experimental): Patient will receive a PEMF treatment. The involved leg will be exposed to PEMF for 10 minutes per session, and the treatment regime will run two times a week for eight weeks, summing up 16 sessions of PEMF exposure in total.
  Interventions: Device: PEMF treatment
- Placebo treatment (Placebo Comparator): Patient will receive a placebo treatment. The involved leg will be exposed to placebo treatment for 10 minutes per session, and the treatment regime will run two times a week for eight weeks, summing up 16 sessions of placebo exposure in total.
  Interventions: Device: Placebo treatment

INTERVENTIONS:
Device: PEMF treatment — Pulsed electromagnetic field (PEMF) therapy is an emerging modality for the treatment of musculoskeletal disorders. Time-varying magnetic pulses are generated by passing an electrical current through a coil. PEMF has been shown to be effective in vitro and in vivo studies for tissue repair and accelerating muscle regeneration. In each treatment, you need to put the reconstructed limb into the machine for 10 minutes.
  Arms: PEMF treatment
Device: Placebo treatment — In this study the placebo group uses the same PEMF machine, but it does not generate any electrical current that have treatment effect. As the active PEMF device does not produce heat or cause any sensation to the tissue, participants are blinded to the treatment. In each treatment, you need to put the reconstructed limb into the machine for 10 minutes.
  Arms: Placebo treatment

SUMMARY:
Anterior cruciate ligament (ACL) tear is common. It accounts for over 50% of all knee injuries. Anterior cruciate ligament reconstruction (ACLR) with hamstring tendon (HT) autograft is the common graft choice for ACLR. However, the outcomes of donor site healing and recovery of muscle strength of HT are not satisfactory, resulting in hamstring muscle weakness and hamstring strength deficit during deep knee flexion, which may lead to hamstring strain after ACLR. Moreover, activation of the hamstring muscle is vital for maintaining dynamic knee joint stability and preventing excessive ACL shear forces. The presence of hamstring muscle deficits after surgery therefore affects the function of the reconstruction ACL. A previous study has reported that the hamstring muscle showed nearly 20% strength deficit at 4 months after ACLR with hamstring autograft

Pulsed electromagnetic field (PEMF) treatment is a non-invasive therapy that has been shown to enhance muscle cell activity and accelerate tissue repair. In clinic, PEMF treatment has been reported to be safe.

This study aims to conduct a double-blinded, placebo-controlled randomised clinical trial to investigate the effects of PEMF therapy for improving the tissue regeneration and strength of the HT donor site in ACLR patients with HT autograft.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female with age ≥ 18 years at the time of surgery
2. First ACLR with HT autograft
3. Both knees without a history of injury/prior surgery
4. LSI for hamstring strength <85% of contralateral leg at 4-month isokinetic assessment (70)
5. Voluntarily agreed to participate and signed the informed consent form

Exclusion Criteria:

1. Any concomitant bone fracture, major meniscus injury or full-thickness chondral injuries requiring altered rehabilitation program post-op
2. Preoperative radiographic signs of arthritis
3. Other associated injuries (fractures and other ligament involvement such as neurovascular bundles injury)
4. Patient with a pacemaker, an implantable defibrillator, neurosurgical clips, a neurostimulator, cochlear implant, a stent, an insulin pump
5. Pregnant or breastfeeding
6. Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Isokinetic Test | Change from baseline (post-ACLR 4 months) hamstring muscle strength at post-ACLR 5 months
  The Cybex dynamometer will be used to test the hamstring muscle strength.
Isokinetic Test | Change from baseline (post-ACLR 4 months) hamstring muscle strength at post-ACLR 6 months
  The Cybex dynamometer will be used to test the hamstring muscle strength.
Isokinetic Test | Change from baseline (post-ACLR 4 months) hamstring muscle strength at post-ACLR 12 months
  The Cybex dynamometer will be used to test the hamstring muscle strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No